CLINICAL TRIAL: NCT02558738
Title: Non Interventional Study (NIS): Clinical Investigation for Evaluation of the Safety and Efficacy of Ectoin Ear Spray and Normison Ear Spray in Skin Treatment of Outer Ear Canal Irritations: A Mulitcenter Non Interventional Study
Brief Title: Non Interventional Clinical Investigation of Ectoin Ear Spray in Skin Treatment of Outer Ear Canal Irritations
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: EOS_PPL-084
Record Dates: First submitted 2015-09-14; First posted 2015-09-24 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pruritus; Dermatitis; Otitis Externa
Keywords: dermatitis and irritations at the outer ear canal; prevention of subacute otitis externa
MeSH Terms: conditions — Pruritus; Dermatitis; Otitis Externa

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Ectoin Ear Spray: treatment according to instruction for use
  Interventions: Device: ear spray
- Normison ear spray: treatment according to instruction for use
  Interventions: Device: ear spray

INTERVENTIONS:
Device: ear spray

SUMMARY:
In this observational study, insights regarding the tolerability and influence on the quality of life of the topical treatment with Ectoin Ear Spray compared to Normison ear spray shall be gained under real life conditions in patients with chronic eczematous irritations and pruritus of the outer ear canal.

ELIGIBILITY:
Inclusion Criteria:

* according to instructions for use

Exclusion Criteria:

* otitis media, acute otitis media
* acute otitis externa
* earache
* perforation of the ear-drum (membrana tympani)
* infections at the ear
* systemic corticosteroid treatment or local at the ear

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care ENT units study the therapeutic process in this observational trial in total of 60 patients in three centres with dermatological irritations of the outer ear canal and pruritus
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pruritus at outer ear canal | 14 days
  assessment of the symptoms on visual analogous scale

SECONDARY OUTCOMES:
Severity of pruritus | 14 days
  assessment of the symptom on Visual Analog Score on values between 0 and 10
Dermatitis | 14 days
  assessment of the symptoms of scaly dermatitis on Visual Analog Score on values between 0 and 10
burning issue on skin | 14 days
  assessment of the symptom on Visual Analog Score on values between 0 and 10
Tolerability: change in VAS score | 14 days
  assessment of tolerability on the Visual Analogue Score on values between 0 and 10
Efficacy: change in VAS score | 14 days
  assessment of efficacy on Visual Analog Score on values between 0 and 10
Change in number of adverse events | 14 days
  incidence of adverse events and correlation to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Sonnemann, Dr med, Principal Investigator — HNO Praxis Elmshorn
Locations (3):
- Germany (3):
  - HNO Praxis Elmshorn, Elmshorn
  - HNO Moeller, Lüneburg
  - HNO Bergmann-Omar, Norderstedt